CLINICAL TRIAL: NCT06277193
Title: Investigation of the Relationship Between Sarcopenia and Balance, Fear of Falling and Fall Risk in Older Female Patients
Status: Completed | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Güreş, Principal Investigator, Doctor, Konya Beyhekim Training and Research Hospital
Other Study IDs: KonyaBeyhekimTRH
Record Dates: First submitted 2024-02-10; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Old; Balance; Fear of falling; Falling risk
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-sarcopenia group: The diagnosis of sarcopenia was determined using EWGSOP2(The European Working Group on Sarcopenia in Older People) criteria. To evaluate walking speed, muscle strength and muscle mass, hand grip test, bioimpedance and 4-meter walking test were performed on each patient, respectively. Those who had results above the critical values determined in muscle strength measurement according to criteria were defined as the group without sarcopenia.
  Interventions: Diagnostic Test: valuation of balance status, fear of falling and risk of falling in patients non-sarcopenia.
- Probable sarcopenia group: Individuals with results below the critical values determined in muscle strength measurement were defined as the probable sarcopenia group if their muscle mass and physical performance values were normal.
  Interventions: Diagnostic Test: Evaluation of balance status, fear of falling and risk of falling in patients with probable sarcopenia.
- Sarcopenia group: If low muscle mass is present in addition to the decrease in muscle strength, this condition is classified as sarcopenia.
  Interventions: Diagnostic Test: Evaluation of balance status, fear of falling and risk of falling in patients with sarcopenia.
- Severe sarcopenia group: If there is a decrease in muscle mass and physical performance along with muscle strength, this condition can be classified as severe sarcopenia.
  Interventions: Diagnostic Test: Evaluation of balance status, fear of falling and risk of falling in patients with severe sarcopenia.

INTERVENTIONS:
Diagnostic Test: valuation of balance status, fear of falling and risk of falling in patients non-sarcopenia. — Daily living activities, frailty, physical performance, balance status, risk of falling, fear of falling, nutritional status, and mental status were evaluated with various scales.
  Groups: Non-sarcopenia group
Diagnostic Test: Evaluation of balance status, fear of falling and risk of falling in patients with probable sarcopenia. — Daily living activities, frailty, physical performance, balance status, risk of falling, fear of falling, nutritional status, and mental status were evaluated with various scales.
  Groups: Probable sarcopenia group
Diagnostic Test: Evaluation of balance status, fear of falling and risk of falling in patients with sarcopenia. — Daily living activities, frailty, physical performance, balance status, risk of falling, fear of falling, nutritional status, and mental status were evaluated with various scales.
  Groups: Sarcopenia group
Diagnostic Test: Evaluation of balance status, fear of falling and risk of falling in patients with severe sarcopenia. — Daily living activities, frailty, physical performance, balance status, risk of falling, fear of falling, nutritional status, and mental status were evaluated with various scales.
  Groups: Severe sarcopenia group

SUMMARY:
This study (study type: cross-sectional) aims to investigate the relationship of sarcopenia level with balance, fear of falling and risk of falling in the elderly female population. In the first stage, 166 participants were divided into two groups: sarcopenia and non-sarcopenia. Afterwards, they were categorized according to sarcopenia level (probable sarcopenia group, sarcopenia group, severe sarcopenia group, group without sarcopenia) and comparisons were made between these subgroups. Then, they were evaluated with various scales and tests (in terms of balance, fear of falling and risk of falling).

DETAILED DESCRIPTION:
The world population is experiencing an aging trend accompanied by declines in fertility and mortality rates. This aging process varies among countries and regions. The aging of societies leads to an increase in health and socioeconomic problems. Sarcopenia is just one of the problems that arise with aging.

Sarcopenia is defined as a progressive syndrome associated with a general loss of muscle mass and strength, leading to a decrease in physical function, deterioration in quality of life, and even adverse outcomes such as death. Although sarcopenia is primarily defined as a syndrome associated with the elderly population, it can also be observed in non-elderly individuals with other diseases or conditions. Therefore, due to its higher prevalence in the elderly population, it can also be referred to as a geriatric syndrome.

The prevalence of sarcopenia varies depending on the measurement methods used to assess muscle mass, muscle strength, and muscle performance, as well as the population studied. The frequency of sarcopenia can range from 8% to 40% in populations aged 60 and over. Muscle mass decreases linearly in both men and women after the age of 40. These losses in muscle mass continue at a rate of 8% per decade up to the age of 70 and increase to 15% in the subsequent decades. Total loss can reach up to 50% in the eighth decade.

The etiology of sarcopenia is multifactorial. Aging, certain chronic diseases, immobility, sedentary lifestyle, and nutritional deficiencies can contribute to sarcopenia. While sarcopenia can sometimes be attributed to a single cause, in most cases, a single cause cannot be identified. Sarcopenia can generally be classified into two main categories: primary and secondary. Primary sarcopenia is solely associated with the aging process, while secondary sarcopenia develops due to one or more causes (such as immobility, comorbidities, nutrition). However, it may not always be possible to make a clear distinction between primary and secondary sarcopenia.

Various imaging methods such as computerized tomography (CT), magnetic resonance imaging (MRI), or dual-energy X-ray absorptiometry (DEXA) can be used to determine muscle mass in the diagnosis of sarcopenia, while anthropometric measurements such as bioimpedance analysis or upper mid-arm circumference and calf circumference may also be applied. Muscle strength is generally measured using a hand dynamometer, while methods such as walking tests, sit-to-stand tests, or stair climbing tests can be used to assess muscle performance.

Individuals who have results below critical values in muscle strength measurement but have normal muscle mass, muscle quality, and physical performance values are defined as probable sarcopenia. If there is also low muscle mass in addition to decreased muscle strength, this condition is classified as sarcopenia. If there is a decrease in muscle mass or quality along with decreased muscle strength and physical performance, this condition can be classified as severe sarcopenia.

Balance is an expression of postural adaptation to changes in the center of gravity during rest or movement. Factors that maintain balance are the integration of vestibular, proprioceptive, and visual data within the central nervous system and coordinated muscle activity resulting from voluntary or involuntary reflex activity. Disruption of balance predisposes to falls. A fall is a condition that usually results in an unwanted change in position, without a significant intrinsic event, strong external force, or intentional movement, usually on the ground or at a lower level. It can also be defined as an uncorrectable change in position.

One of the psychological consequences of falling is fear of falling. This is defined as an anxiety condition that leads to avoidance of physical activity after a fall. This condition is often accompanied by anxiety and loss of confidence. Fear of falling may decrease over time or become continuous. Previous fall events, advanced age, being female, vision problems, depressive mood, polypharmacy, and balance disorders can be among the risk factors for fear of falling.

Studies have found that sarcopenia is associated with many diseases, reduces quality of life, increases dependency, affects mortality, and increases hospitalizations. However, studies investigating the relationship between balance, risk of falling, fear of falling, and sarcopenia are limited in the literature. This study aims to investigate the relationship between the level of sarcopenia and balance, fear of falling, and risk of falling in an elderly female population.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 60 years old
2. Being a woman

Exclusion Criteria:

1. Those under 60 years of age
2. Male ones
3. Hand deformities
4. Advanced knee osteoarthritis
5. Advanced hand osteoarthritis
6. Advanced osteoarthritis in the waist and hip area
7. History of Carpal Tunnel Syndrome
8. Communication disorders
9. Muscle diseases
10. Root compressions
11. History of upper and lower extremity spine surgery, prostheses and previous fracture history
12. Those with advanced kyphosis and scoliosis
13. Those with serious neck problems
14. Lumbar spinal stenosis
15. Those with decompensated heart, liver and kidney failure
16. Those who have any disease (neurological, orthopedic, metabolic, etc.) that causes balance disorders
17. Those who use medication that may cause balance disorders
18. Those with severe hearing and vision impairment
19. History of antidepressant, anticholinergic, benzodiazepine and anxiolytic use in the last 3 months
20. Those with major psychiatric illness
21. Those who use alcohol regularly
22. Patients with pacemakers
23. Those with immobility, those whose mobilization is limited for some reason

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 208 patients who applied to the outpatient clinic were examined for eligibility for the study. During the detailed evaluation process, patients who did not meet the exclusion criteria (communication problems, etc.) and did not want to participate in the study were excluded from the study. Detailed histories were taken from the remaining 166 participants and physical examinations were performed.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Sociodemographic data | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  A form was created to determine the sociodemographic characteristics of the patients. In addition, data on the number of falls and fractures in the last year was also obtained in this form.
Berg Balance Scale(BBS) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  The Berg balance scale was initially developed to evaluate postural control and is now widely used in many fields. Scoring is done on a 5-point scale that evaluates whether the patient can perform the task safely and independently within a certain period of time. 0 points are given for unrealizable performances and 4 points are given for normal performances. The points given are added together to obtain the maximum score. 0-20 points indicate high fall risk, 21-40 points indicate medium fall risk, 41-56 points indicate low fall risk.
Falls Efficacy Scale (FES) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  Developed based on low perceived self-efficacy, FES is a reliable and valid method to measure fear of falling. Such as taking a bath, taking a shower, reaching shelves, walking around the house, preparing meals without carrying heavy or hot objects, getting in and out of bed, answering the door or telephone ring, sitting on a chair and getting up, dressing and undressing, going to the toilet and leaving the toilet, personal care. Patients are asked to rate their daily living activities. The points given are evaluated between "1 point I trust very much" and "10 points I do not trust at all", the scores between 0 and 10 are summed and the resulting score is recorded.
Balance and Gait Assessment Scale | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  This scale is an important tool to evaluate the individual's functional status and daily living activities. The scale consists of a maximum of 16 points for balance and a maximum of 12 points for walking, for a total of 28 points. Individuals who score 26 or below on the scale are thought to have a problem; For those with scores of 19 or below, it is observed that the risk of self-falling increases fivefold compared to normal individuals.

SECONDARY OUTCOMES:
Biochemical data | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  The most current biochemical data in the hospital system within the last year were recorded.
Co-morbidities | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  Comorbidities of the patients were recorded.(like hypertension, heart disease...etc.)
Number of drugs | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  Medications used due to comorbidities were questioned.
Basic activities of daily living (Katz) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  The ADL Index, developed by Katz and his team in 1963, determines activities aimed at fulfilling the basic needs for the continuation of life. The ADL Index includes six questions about bathing, dressing, toileting, movement, excretion and feeding activities. Scoring is made between 0 and 6, and an increase in the score is associated with an increase in the level of independence.
Instrumental activities of living (Lawton-Brody; IADL) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  Developed by Lawton and Brody in 1969, IADL determines the instrumental daily living activities of individuals. The IADL Index includes eight questions about using the phone, preparing meals, shopping, doing daily household chores, doing laundry, taking transportation, using medications, and money management. Scoring is made between 0 and 8, and the increase in the score is related to the increase in the level of independence.
Mini-nutritional evaluation (MNA-Short form) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  Mini-nutritional assessment-short form consists of six items that have been determined to have a high correlation with conventional nutritional assessment. In this evaluation, scoring is done by looking at factors such as the change in the patient's appetite, whether there has been weight loss in the last three months, mobility, whether the patient has experienced psychological distress or acute illness in the last three months, the presence of neuropsychological problems and body mass index.
Mini-mental state assessment (MMSE) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  Folstein et al. Developed in 1975, this brief screening test is the most commonly used test for dementia screening. It consists of eleven questions and is evaluated out of 30 points. Scores between twenty-four and thirty points may reflect normal, scores between 18-23 points may reflect mild dementia, and scores of 17 points and below may reflect severe dementia. This test evaluates areas such as orientation, memory, attention, calculation, recall, language, motor function and perception, and its biggest advantage is that it can be easily and quickly applied.
Yesavage Geriatric Depression Scale Short Form (GDS-SF) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  GDS-SF, developed by Yesavage et al. in 1983, is used to screen for depression in elderly patients. The 15-question short form, developed by Burke et al. in 1991 and proven to be valid and reliable, is preferred for its ease of use. GDS-SF is a screening test that can be applied quickly and easily. Scores of five points and above may be compatible with depression, but the patient's clinical condition should also be taken into account for a definitive assessment. This test provides an advantage in that it can be applied to patients with dementia.
FRAIL fragility index | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  The "FRAIL Scale", developed by Morley and his team in 2012, is an evaluation tool consisting of 5 items. This scale receives a score of 0 or 1 for each item, depending on the answers given by the patients. As a result of the total scoring, those who score 0 points are classified as "non-frail", those who score 1-2 points are classified as "pre-frail", and those who score more than 2 points are classified as "frail".
Short physical performance battery (SPPB) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  SPPB was used to evaluate physical function. SPPB includes 3 objective tests that evaluate lower extremity function; Walking 4 meters, getting up from a chair and standing balance. The total test score ranges from 0 to 12. High scores indicate strong lower extremity function and a low risk of falling
Timed up and go test (TUG) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  A short, simple and reliable test used to evaluate balance function involves tasks such as getting up from a chair, walking 3 meters forward, turning 180 degrees in place, walking back to the chair and sitting down. While the person performs these tasks, time is kept with a stopwatch. There is a significant relationship between the time to complete the test and the level of functional mobility. It was observed that people who completed the test in less than 20 seconds were independent in transfer, received high scores on BBS, and achieved the required walking speed (0.5 m/sec) in society. It was determined that people who completed the test in 30 seconds or more were more dependent on their daily living activities, needed assistive devices for ambulation, and had lower scores on BBS.
The Tampa Scale for Kinesiophobia (TSK) | During the initial evaluation of the patients, their information was recorded in approximately 1 hour.
  TSK was originally developed in 1991 but was not published. This original scale was later republished in 1995 with the permission of the researchers who developed it. TSK is a 17-item scale designed to measure fear of movement-related injury. The scale includes fear-avoidance parameters in cases of injury or re-injury in work-related activities.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih güreş, Principal Investigator — assistant doctor
Locations (1):
- Konya Beyhekim Training and Research Hospital Physical Medicine and Rehabilitation Clinic, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Batsis JA, Buscemi S. Sarcopenia, sarcopenic obesity and insulin resistance. Medical Complications of Type 2 Diabetes: IntechOpen; 2011. p. 233-56
- [Background] Abellan van Kan G. Epidemiology and consequences of sarcopenia. J Nutr Health Aging. 2009 Oct;13(8):708-12. doi: 10.1007/s12603-009-0201-z. PMID 19657554
- [Background] Metter EJ, Conwit R, Tobin J, Fozard JL. Age-associated loss of power and strength in the upper extremities in women and men. J Gerontol A Biol Sci Med Sci. 1997 Sep;52(5):B267-76. doi: 10.1093/gerona/52a.5.b267. PMID 9310077
- [Background] Rolland Y, Lauwers-Cances V, Cournot M, Nourhashemi F, Reynish W, Riviere D, Vellas B, Grandjean H. Sarcopenia, calf circumference, and physical function of elderly women: a cross-sectional study. J Am Geriatr Soc. 2003 Aug;51(8):1120-4. doi: 10.1046/j.1532-5415.2003.51362.x. PMID 12890076
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] ŞAHİN G, ŞEKER H, YEŞİLIRMAK M, ÇADIR A. Denge diski egzersizlerinin dinamik denge ve duruş kontrolü üzerindeki etkisinin incelenmesi. Spor ve performans araştırmaları dergisi. 2015;6(1):50-7.
- [Background] Alkan S. 65 yaş ve üstü bireylerde D vitamini düzeyi ile düşme riski arasındaki ilişki. 2009.
- [Background] Akman MN, Karataş M. Temel ve uygulanan kinezyoloji: Haberal Eğitim Vakfı; 2003.
- [Background] Stel VS, Smit JH, Pluijm SM, Lips P. Balance and mobility performance as treatable risk factors for recurrent falling in older persons. J Clin Epidemiol. 2003 Jul;56(7):659-68. doi: 10.1016/s0895-4356(03)00082-9. PMID 12921935
- [Background] ÇINARLI T, Zeliha K. 65 Yaş Ve Üzeri Yaşlılarda Düşme Risk Ve Korkusunun Günlük Yaşam Aktiviteleri Ve Yaşam Kalitesi Üzerine Etkisi. Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi. 2015;4(4):660-79.
- [Background] Tinetti ME, Williams TF, Mayewski R. Fall risk index for elderly patients based on number of chronic disabilities. Am J Med. 1986 Mar;80(3):429-34. doi: 10.1016/0002-9343(86)90717-5. PMID 3953620
- [Background] Schepens S, Sen A, Painter JA, Murphy SL. Relationship between fall-related efficacy and activity engagement in community-dwelling older adults: a meta-analytic review. Am J Occup Ther. 2012 Mar-Apr;66(2):137-48. doi: 10.5014/ajot.2012.001156. PMID 22394523
- [Background] Carpenter CR. Evidence-based emergency medicine/systematic review abstract. Preventing falls in community-dwelling older adults. Ann Emerg Med. 2010 Mar;55(3):296-8. doi: 10.1016/j.annemergmed.2009.06.014. Epub 2009 Jul 17. No abstract available. PMID 19615786
- [Background] Oh-Park M, Xue X, Holtzer R, Verghese J. Transient versus persistent fear of falling in community-dwelling older adults: incidence and risk factors. J Am Geriatr Soc. 2011 Jul;59(7):1225-31. doi: 10.1111/j.1532-5415.2011.03475.x. Epub 2011 Jun 30. PMID 21718266
- [Background] Cawthon PM, Marshall LM, Michael Y, Dam TT, Ensrud KE, Barrett-Connor E, Orwoll ES; Osteoporotic Fractures in Men Research Group. Frailty in older men: prevalence, progression, and relationship with mortality. J Am Geriatr Soc. 2007 Aug;55(8):1216-23. doi: 10.1111/j.1532-5415.2007.01259.x. PMID 17661960
- [Background] Cawthon PM, Fox KM, Gandra SR, Delmonico MJ, Chiou CF, Anthony MS, Sewall A, Goodpaster B, Satterfield S, Cummings SR, Harris TB; Health, Aging and Body Composition Study. Do muscle mass, muscle density, strength, and physical function similarly influence risk of hospitalization in older adults? J Am Geriatr Soc. 2009 Aug;57(8):1411-9. doi: 10.1111/j.1532-5415.2009.02366.x. PMID 19682143